CLINICAL TRIAL: NCT05443711
Title: SARCOBEAGING: Sarcopenic Obesity as a Risk of Premature Aging
Brief Title: Sarcopenic Obesity as a Risk of Premature Aging
Acronym: SARCOBEAGING
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital de Leon (Other Government)
Collaborators: Universidad de León (Other)
Responsible Party: Principal Investigator, Maria D. Ballesteros Pomar, Head of Clinical Nutrition Unit, Endocrinology and Nutrition, Hospital de Leon
Other Study IDs: CAULE 21125; GRS 2326/A/21 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y León)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Sarcopenic Obesity; Aging
Keywords: obesity; sarcopenia; aging; klotho; miRNA
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obesity: Patients with obesity attended in the High-Risk Obesity clinic of the Complejo ASistencial Universitario de León, 50-60 years-old
  Interventions: Other: No intervention, observational study
- control: control group of healthy people of the same age group without obesity or cardiovascular risk factors that will be selected among volunteers from the CAULE staff. and University of Leon
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — No intervention, observational study

SUMMARY:
Recently, numerous signaling proteins derived from adipose tissue and/or skeletal muscle have been described and are involved in the pathogenesis of obesity and the pathophysiology of aging. Current evidence suggests a role for the FGF-Klotho system, circulating cell-free DNA (cfDNA), miR-499, and exosomes not only in the pathophysiology of obesity, but also in the association with sarcopenic obesity (OS) and in a accelerated aging.

The investigator´s hypothesis is that obesity, especially OS, might be the cause of advanced aging, reflected in lower levels of the FGF-Klotho system, higher concentrations of cfDNA and a change in the profiles of miRNAs and exosomes, which could have an impact on risk. cardiovascular and metabolic.

For this, a descriptive cross-sectional study is proposed in 50 patients with obesity, who will be classified as OS or not, and 25 healthy controls, between 50-60 years old. The determinations are made by the IBIOMED of the University of León.

To study the evolution of aging markers over a year of follow-up, a second part of the study will analyze the possible differences according to the treatments assigned to each patient in the context of real life (lifestyle changes, drugs, bariatric surgery).

DETAILED DESCRIPTION:
Descriptive cross-sectional study in patients with obesity attended in the High-Risk Obesity consultation of the University Assistance Complex of León, with a control group of healthy people of the same age group without obesity or cardiovascular risk factors that will be selected among volunteers from the CAULE and University of Leon staff.

The second part of the study will be a one-year prospective longitudinal follow-up study of the patients included in the first part of the study.

ELIGIBILITY:
Inclusion Criteria:

* People, men and postmenopausal women, aged between 50 and 60 years. Diagnosis of central obesity with body mass index greater than or equal to 30 kg/m2 and waist circumference equal to or greater than 102 cm in men and 88 cm in women.

Control group, of healthy individuals with BMI less than 30 kg/m2 and waist circumference <102 cm in men and <88 cm in women, of the same age group and matched according to gender.

Able of giving informed consent.

Exclusion Criteria:

* Premenopausal women. Kidney disease with glomerular filtration rate less than 60. Liver disease with plasma GOT/GPT/GGT levels greater than x 2 the upper limit of normal.

Active cancer disease. Heart or respiratory failure requiring pharmacological treatment.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People, men and postmenopausal women, aged between 50 and 60 years. Diagnosis of central obesity with body mass index greater than or equal to 30 kg/m2 and waist circumference equal to or greater than 102 cm in men and 88 cm in women.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
S-Klotho levels | 2022-2023
miR-499 | 2022-2023
  Blood samples
cfDNA | 2022-2023
  Blood samples
Exosomes | 2022-2023
  Blood samples

SECONDARY OUTCOMES:
Fat mass | 2022-2023
  DXA
Muscle mass | 2022-2023
  DXA
Muscle function | 2022-2023
  Hand grip strength
Muscle function 2 | 2022-2023
  Strenght platform

CONTACTS AND LOCATIONS:
Overall Officials: Maria D Ballesteros Pomar, PhD, Study Director — Complejo Asistencial Universitario de León
Locations (1):
- Complejo Asistencial Universitario de León, León, Spain

IPD SHARING:
Plan to Share IPD: No